CLINICAL TRIAL: NCT04689672
Title: Predictivity of hEmoGasAnalysis Associated to Bedside Lung UltraSound in Determining COVID-19 Severity in the Emergency Departement
Brief Title: Predictivity of Hemogasanalysis and Lung UltraSound in Determining COVID-19 Severity
Acronym: COVID-PEGALUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paola Maffi, Associate Professor in Internal Medicine; Head of School of Emergency Medicine, IRCCS San Raffaele
Other Study IDs: COVID-PEGALUS
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Bedside lung ultrasound

SUMMARY:
This retrospective-prospective longitudinal observational study was designed to evaluate the role of bedside lung ultrasound per se and in association with hemogasanalysis parameters in predicting the severity of COVID-19 patients in the Emergency Departement (ED).

Retrospective data regarding patients who presented at the ED of IRCCS San Raffaele Hospital from 10/11/2020, together with those acquired by the observation of patients who will access to the ED until 10/05/2021 will be collected, configuring a total enrollment period of 6 months.

Clinical informations about patients' medical history will be recorded, with particular focus on the type and date of onset of the symptoms. The diagnostic and therapeutic strategy will be chosen according to the current standard of care. Results of bedside lung ultrasound, together with vital parameters, blood gas analysis, laboratory and other findings will be recorded.

The primary outcome will be defined as patients' outcome at time of discharge from the ED, in terms of intensity of required care (home discharge, low or high-intensity care hospitalization, death). Secondary outcomes will be patients' prognosis 30 days after access to ED and the required intensity of care (eg need for non-invasive ventilation, oro-tracheal intubation).The follow-up 30 days after access to the ED will be evaluated by telephone survey or by consulting medical records.

ELIGIBILITY:
Inclusion Criteria:

* SARS - CoV 2 infection confirmed by positive RT-PCR on nasopharyngeal swab

Exclusion Criteria:

* impossibility to perform lung ultrasound due to technical limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to IRCCS San Raffaele Hospital Emergency Departement with SARS CoV-2 documented infection from 10/11/2020 to 10/05/2021.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
Patients' short-term outcome | Up to 7 days
  Patients' outcome at time of discharge from the Emergency Departement, expressed in terms of intensity of required care (home discharge, low or high-intensity care hospitalization, death).

SECONDARY OUTCOMES:
Patients' long-term outcome | 30 days after access to the Emergency Departement
  Patients' outcome 30 days after access to the Emergency Departement, expressed in terms of intensity of required care (home discharge, low or high-intensity care hospitalization, death).
Intensity of care | Up to 7 days
  Required intensity of care during the observational period in the Emergency Departement (eg need for non-invasive ventilation, oro-tracheal intubation).

CONTACTS AND LOCATIONS:
Overall Officials: Paola AM Maffi, MD, PhD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

REFERENCES:
- [Result] Khalili N, Haseli S, Iranpour P. Lung Ultrasound in COVID-19 Pneumonia: Prospects and Limitations. Acad Radiol. 2020 Jul;27(7):1044-1045. doi: 10.1016/j.acra.2020.04.032. Epub 2020 May 3. No abstract available. PMID 32444253
- [Result] Smith MJ, Hayward SA, Innes SM, Miller ASC. Point-of-care lung ultrasound in patients with COVID-19 - a narrative review. Anaesthesia. 2020 Aug;75(8):1096-1104. doi: 10.1111/anae.15082. Epub 2020 Apr 28. PMID 32275766
- [Result] Lu X, Zhang M, Qian A, Tang L, Xu S. Lung ultrasound score in establishing the timing of intubation in COVID-19 interstitial pneumonia: A preliminary retrospective observational study. PLoS One. 2020 Sep 3;15(9):e0238679. doi: 10.1371/journal.pone.0238679. eCollection 2020. PMID 32881950 (Retraction: PMID 33382851 PLoS One. 2020 Dec 31;15(12):e0245032)
- [Result] Manivel V, Lesnewski A, Shamim S, Carbonatto G, Govindan T. CLUE: COVID-19 lung ultrasound in emergency department. Emerg Med Australas. 2020 Aug;32(4):694-696. doi: 10.1111/1742-6723.13546. Epub 2020 Jun 16. PMID 32386264
- [Result] Dargent A, Chatelain E, Kreitmann L, Quenot JP, Cour M, Argaud L; COVID-LUS study group. Lung ultrasound score to monitor COVID-19 pneumonia progression in patients with ARDS. PLoS One. 2020 Jul 21;15(7):e0236312. doi: 10.1371/journal.pone.0236312. eCollection 2020. PMID 32692769